CLINICAL TRIAL: NCT00996021
Title: A Study to Evaluate the Effect of a Single 250 mg Oral Dose of GSK1349572 on Cardiac Conduction as Assessed by 12-lead Electrocardiogram Compared to Placebo and a Single Oral Dose of Moxifloxacin (ING111856).
Brief Title: Study to Assess Cardiac Conduction of GSK1349572
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 111856
Record Dates: First submitted 2009-10-08; First posted 2009-10-16 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Healthy Subjects
Keywords: GSK1349572; moxifloxacin; Avelox; QTc
MeSH Terms: interventions — dolutegravir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Arm 1 (Experimental): This is a three way crossover study with 3 periods. Subjects will receive a single dose of either GSK1349572 250 mg suspension, placebo suspension or moxifloxacin 400 mg tablet in each of the three periods. The order in which the treatments are given will be randomized. There is a screening visit within 30 days prior to the first dose of study drug and a follow-up visit within 10-14 days after the last dose of study drug.
  Interventions: Drug: GSK1349572 250 mg; Drug: Placebo Suspension; Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: GSK1349572 250 mg — This is an experimental HIV medication in the integrase inhibitor class.
Drug: Placebo Suspension — Placebo is a liquid with no drug in it.
Drug: Moxifloxacin 400 mg — This is an FDA approved antibiotic in the fluoroquinolone class.
  Other Names: AVELOX. AVELOX is a registered trademark of Bayer Aktiengesellschaft

SUMMARY:
This will be a randomized, partial-blind, placebo-controlled, single dose, cross-over trial investigating the effect of GSK1349572 on cardiac repolarization as compared to placebo in healthy adult males and females. Approximately 42 subjects will be enrolled in this study and will be admitted to the clinic for three separate dosing sessions. Subjects will receive single dose administrations of placebo, a supratherapeutic dose of GSK1349572 (250 mg), and moxifloxacin (400 mg) in random sequence. Safety of subjects will be monitored by clinical observation, measures of vital signs, 12-lead ECGs and clinical laboratory measurements.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [or Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 3 days after the last dose of study drug.
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to the first dose of study medication.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, inflammatory bowel disease or pancreatitis should be excluded.
* Subjects with active peptic ulcer disease.
* Subjects with a history of upper gastrointestinal bleeding,
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease. Personal or family history of long QT syndrome.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatobiliary diseases. Subjects with a history of nephrolithiasis will be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of 2nd degree or higher AV block.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Subjects with a hemoglobin <12 g/dL.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* ECG within protocol limits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF for GSK1349572. | 24 hours

SECONDARY OUTCOMES:
Safety and tolerability of GSK1349572 as assessed by 12-lead ECGs, vital signs, adverse events, and clinical laboratory tests. | 24 hours
Change from baseline in QTcB, QTci, QT, and HR for GSK1349572 | 24 hours
Change from baseline in QTcF, QTcB, QTci, QT, and HR for placebo | 24 hours
Change from baseline in QTcF, QTcB, QTci, QT, and HR for moxifloxacin | 24 hours
AUC(0-24), AUC(0-t), AUC(0-tau), Cmax, tmax, CL/F, Vdz/F, and t1/2 from plasma concentrations of GSK1349572 and moxifloxacin (if needed) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States